CLINICAL TRIAL: NCT06417931
Title: A Pharmacist-Led Intervention on Medication Adherence and Inhaler Usage on Clinical Outcomes Among Patients With Asthma and Chronic Obstructive Pulmonary Disease in Ibadan, Nigeria
Brief Title: Medication Adherence and Use of Inhaler Devices in Patients With Asthma or COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ibadan (Other)
Responsible Party: Principal Investigator, Uyiose Fortress Ufuah, Graduate Student, University of Ibadan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Medication adherence
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Asthma COPD
MeSH Terms: interventions — Patient Education as Topic; Counseling

STUDY DESIGN:
Intervention Model Description: Quasi-randomised control trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental): Patients in the intervention group received education and counselling tips about their disease condition and medications
  Interventions: Behavioral: Patient education and counselling

INTERVENTIONS:
Behavioral: Patient education and counselling — The pharmacist intervention was aimed at identifying and addressing barriers to treatment adherence through tailored strategies
  Arms: Intervention

SUMMARY:
This study aims to evaluate the impact of a pharmacist-led intervention programme on medication adherence and use of inhaler devices on clinical outcomes of patients with asthma and COPD attending a tertiary health facility in Nigeria.

DETAILED DESCRIPTION:
Medication non-adherence in asthma and COPD patients have been established to be very high, and along-side poor knowledge of proper use of inhaler devices, results in suboptimal disease control among these patients. Studies evaluating the impact of a comprehensive intervention on medication adherence and inhaler usage on disease control are scare in developing countries. This study was a prospective single-blind quasi-randomized-controlled study among asthma and COPD patients attending the chest out-patient clinic of the University College Hospital, Ibadan. The baseline questionnaire was administered to consenting patients to explore demographic and specific clinical characteristics, knowledge of the disease, current medications, medication adherence, knowledge of use of metered dose (MDIs) and diskus inhalers, and asthma/COPD control status using the asthma control test (ACT) and COPD assessment test (CAT) scales. Subsequently, patients were assigned into intervention or control groups using odd or even number assignation. Patients in the intervention group were followed up for two months via face to face interviews, short message services, and phone calls at one-weekly intervals, so as to provide education and counseling to resolve the identified gaps during the baseline interaction. Descriptive statistics were used to summarize the data, while chi-square, t-test, Fishers exact test and Wilcoxon-signed ranked tests were used as appropriate to test for associations at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

Patients 18 years of age and older with a primary diagnosis of asthma or COPD by a physician who are willing to complete the study and have telephone access

Exclusion Criteria:

All non-consenting patients and patients who are not on any medications at any point in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Medication adherence | Two months
  The difference between the intervention and control groups with respect to the changes in the medication adherence score from baseline to a 2-month follow-up.
Use of inhaler devices | Two months
  The difference between the intervention and control groups with respect to the changes in knowledge of the use of inhaler devices from baseline to a 2-month follow-up.

SECONDARY OUTCOMES:
disease control | Two months
  The difference in asthma or Chronic obstructive pulmonary disease (COPD) control among patients in control and intervention groups from baseline to 2-months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- University College Hospital, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adisa R, Ufuah UF, Ige OM. Impact of pharmacist-led intervention in medication adherence and inhaler usage on asthma and chronic obstructive pulmonary disease control: a quasi-experimental study. BMC Health Serv Res. 2024 Oct 8;24(1):1199. doi: 10.1186/s12913-024-11683-9. PMID 39379970